CLINICAL TRIAL: NCT00264576
Title: A Phase 2, Observer-Blinded, Randomized, Multicenter Study in Healthy Adults to Evaluate Safety and Tolerability and to Compare Immunogenicity of a Single Dose of Either an Investigational Trivalent Inactivated Influenza Vaccine Produced in Mammalian Cell Culture or a US-licensed Trivalent Inactivated Influenza Vaccine (Fluvirin®) Produced in Embryonated Hen Eggs
Brief Title: Study of the Safety and Immunogenicity of an Influenza Vaccine Administered to Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Collaborators: Novartis Vaccines and Diagnostics (formerly Chiron Vaccines) (Unknown)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V58P5
Record Dates: First submitted 2005-12-09; First posted 2005-12-13 (Estimated); Results first posted 2013-01-28 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2012-12

CONDITIONS: Influenza Disease; Flu
Keywords: influenza; flu
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- cTIV (Experimental): Received one dose of cell-culture derived trivalent influenza vaccine (cTIV).
  Interventions: Biological: Influenza Virus Vaccine
- TIV (Active Comparator): Received one dose of egg-derived trivalent vaccine (TIV).
  Interventions: Biological: Influenza Virus Vaccine

INTERVENTIONS:
Biological: Influenza Virus Vaccine

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of cell culture-derived, inactivated, subunit influenza vaccine in comparison to licensed Fluvirin vaccine administered to healthy adults ages 18 < 50 years.

ELIGIBILITY:
Inclusion Criteria:

18 to <50 years of age;

1. able to comprehend and follow all required study procedures;
2. able and willing to provide written informed consent prior to study entry;
3. available for all the visits scheduled in the study;
4. in general good health as determined by:

   1. subject-reported medical history,
   2. physical examination by a qualified study nurse, a physician's assistant, or a physician,
   3. clinical judgment of the investigator; among all female volunteers, evidence of a negative pregnancy test conducted on the same day as and prior to study vaccination, and agreement to practice adequate contraception for at least 6 weeks after vaccination as further described in the protocol.

Exclusion Criteria:

1. received influenza vaccine within the past 6 months;
2. laboratory-confirmed influenza disease in the past 6 months;
3. any acute respiratory disease or infection requiring systemic antibiotic or antiviral therapy (chronic antibiotic therapy for urinary tract prophylaxis was acceptable) or fever ≥38°C (100.4°F) within the past 3 days;
4. receipt of another investigational agent within 90 days or before completion of the safety follow-up period in another study, whichever was longer, prior to enrollment, and unwilling to refuse participation in another investigational study through the end of the study;
5. any history of or current serious disease, such as: d) cancer (except for benign or localized skin cancer), e) autoimmune disease (including rheumatoid arthritis), f) advanced arteriosclerotic disease or diabetes mellitus, g) chronic obstructive pulmonary disease (COPD), h) acute, chronic, or progressive hepatic disease, i) acute, chronic, or progressive renal disease, j) congestive heart failure, k) bleeding diathesis, l) an inherited genetic anomaly (known cytogenic disorders, e.g., Down's Syndrome), m) any other serious, acute, or chronic disease including progressive neurological disease or seizure disorder unrelated to fever;
6. surgery or hospitalization planned during the study period;
7. history of any anaphylaxis, serious vaccine reactions, vaccine-associated oculorespiratory syndrome, or allergy to eggs, egg products, mercury-containing compounds (such as sodium-ethyl-mercuro-thio-salicylate), or any other vaccine component or component of the potential packaging materials (latex);
8. known or suspected disease of the immune system, or receiving immunosuppressive therapy, including use of: n) systemic corticosteroids, known to be associated with suppression of the hypothalamic-pituitary-adrenal (HPA) axis (i.e., systemic corticosteroids [15 mg/day of prednisone or its equivalent] or chronic use of inhaled high potency corticosteroids [budesonide 800 μg/day or fluticasone 750 μg/day]), both within the previous 60 days, o) receipt of immunostimulants within 60 days, p) receipt of parenteral immunoglobulin preparation, blood products, and/or plasma derivatives within the 3 months prior to study entry or anticipated during the full length of the study;
9. at high risk for developing an immunocompromising disease;
10. history of (or current) drug or alcohol abuse that in the investigator's opinion would interfere with safety of the subject or the evaluation of study objectives;
11. pregnant or breastfeeding;
12. if female of childbearing potential, refusal to use a reliable contraceptive method, as described further in the protocol, during the first 6 weeks after vaccination;
13. if female of childbearing potential and sexually active, has not used any of the following birth control methods for the specified time period prior to study entry:

    1. hormonal (e.g., oral, injection, transdermal patch, implant, cervical ring), barrier (e.g., condom with spermicide or diaphragm with spermicide), or intrauterine device (e.g., IUD) for 2 months or more prior to study entry,
    2. monogamous relationship with vasectomized partner: partner has been vasectomized for 6 months or more prior to the subject's study entry;
14. obese (e.g., with a body mass index [BMI] ≥35, where BMI reflects obesity and not high muscle mass);
15. any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives or might interfere with the safety of the study subject.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 613 (Actual)
Dates: Start 2005-10; Primary Completion 2005-12 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (3):
- United States (3):
  - Bardstown, Kentucky
  - Pittsburgh, Pennsylvania
  - Salt Lake City, Utah

REFERENCES:
- [Result] Reisinger KS, Block SL, Izu A, Groth N, Holmes SJ. Subunit influenza vaccines produced from cell culture or in embryonated chicken eggs: comparison of safety, reactogenicity, and immunogenicity. J Infect Dis. 2009 Sep 15;200(6):849-57. doi: 10.1086/605506. PMID 19673652

RESULTS

PARTICIPANT FLOW:
Groups:
- cTIV: Adults 18 to < 50 years of age received one dose of cell-culture-derived trivalent influenza vaccine (cTIV).
- eTIV_f: Adults 18 to < 50 years of age received one dose of egg-derived trivalent vaccine (eTIV_f).
Period: Overall Study
Arm/Group | cTIV | eTIV_f
Started | 308 | 305
Completed | 307 | 304
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | cTIV | eTIV_f | Total
Number analyzed (Participants) | 308 | 305 | 613
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (8.8) | 34.2 (9.3) | 34 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196 | 205 | 401
  Male | 112 | 100 | 212

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMT) After 1 Dose of Cell-culture-derived Vaccine (cTIV) or Egg-derived Vaccine (eTIV_f), Using the ANOVA Method.
Description: Non-inferiority was measured by the ratio of postvaccination geometric mean titers (cTIV vs. eTIV_f) against all three vaccine strains as assessed by egg-derived antigen and cell-derived antigen haemagglutination inhibition (HI) assay.
Time Frame: 3 weeks postvaccination (Day 22)
Population: Analysis was done on per protocol set
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | cTIV | eTIV_f
Number analyzed (Participants) | 307 | 303
Titer
  A/H1N1 (egg-derived assay) | 259 [225 to 298] | 306 [265 to 352]
  A/H3N2 (egg-derived assay) | 181 [157 to 210] | 320 [276 to 370]
  B (egg-derived assay) | 179 [157 to 203] | 157 [138 to 179]
  A/H1N1 (cell-culture-derived assay) | 468 [407 to 538] | 508 [441 to 585]
  A/H3N2 (cell-culture-derived assay) | 287 [250 to 331] | 468 [406 to 539]
  B (cell-culture-derived assay) | 176 [155 to 199] | 134 [118 to 153]
Statistical Analysis 1: Comparison: cTIV vs eTIV_f; The following hypotheses were tested for A/H1N1 strain as measured by HI egg-derived assay: H0i: log(GMTeTIV_f(i)) - log(GMTcTIV(i)) ≥0.301 ↔ GMTcTIV(i) / GMTeTIV_f(i) ≤0.5 (null hypothesis); H1i: log(GMTeTIV_f(i)) - log(GMTcTIV(i)) <0.301 ↔ GMTcTIV(i) / GMTeTIV_f(i) >0.5 (alternative hypothesis); With: GMTcTIV(i)=GMT for strain i in cTIV group; GMTeTIV_f(i)=GMT for strain i in eTIV_f group; Test type: Non-Inferiority or Equivalence — To demonstrate non-inferiority of cTIV to eTIV_f the lower limit of the 95% confidence interval (CI) around the ratio of the postvaccination GMTs had to be >0.5; ANOVA; Ratio of GMT = 0.85, 95% CI 2-sided [0.70 to 1.04]
Statistical Analysis 2: Comparison: cTIV vs eTIV_f; The following hypotheses were tested for A/H3N2 strain as measured by HI egg-derived assay: H0i: log(GMTeTIV_f(i)) - log(GMTcTIV(i)) ≥0.301 ↔ GMTcTIV(i) / GMTeTIV_f(i) ≤0.5 (null hypothesis); H1i: log(GMTeTIV_f(i)) - log(GMTcTIV(i)) <0.301 ↔ GMTcTIV(i) / GMTeTIV_f(i) >0.5 (alternative hypothesis); With: GMTcTIV(i)=GMT for strain i in cTIV group; GMTeTIV_f(i)=GMT for strain i in eTIV_f group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Ratio of GMT = 0.57, 95% CI 2-sided [0.46 to 0.70]
Statistical Analysis 3: Comparison: cTIV vs eTIV_f; The following hypotheses were tested for B strain as measured by HI egg-derived assay: H0i: log(GMTeTIV_f(i)) - log(GMTcTIV(i)) ≥0.301 ↔ GMTcTIV(i) / GMTeTIV_f(i) ≤0.5 (null hypothesis); H1i: log(GMTeTIV_f(i)) - log(GMTcTIV(i)) <0.301 ↔ GMTcTIV(i) / GMTeTIV_f(i) >0.5 (alternative hypothesis); With: GMTcTIV(i)=GMT for strain i in cTIV group; GMTeTIV_f(i)=GMT for strain i in eTIV_f group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Ratio of GMT = 1.14, 95% CI 2-sided [0.95 to 1.36]
Statistical Analysis 4: Comparison: cTIV vs eTIV_f; The following hypotheses were tested for A/H1N1 strain as measured by HI cell-culture-derived assay: H0i: log(GMTeTIV_f(i)) - log(GMTcTIV(i)) ≥0.301 ↔ GMTcTIV(i) / GMTeTIV_f(i) ≤0.5 (null hypothesis); H1i: log(GMTeTIV_f(i)) - log(GMTcTIV(i)) <0.301 ↔ GMTcTIV(i) / GMTeTIV_f(i) >0.5 (alternative hypothesis); With: GMTcTIV(i)=GMT for strain i in cTIV group; GMTeTIV_f(i)=GMT for strain i in eTIV_f group; Test type: Non-Inferiority or Equivalence — To demonstrate non-inferiority of cTIV to eTIV_f the lower limit of the 95% confidence interval (CI) around the ratio of the postvaccination geometric mean titers (GMTs) had to be >0.5; ANOVA; Ratio of GMT = 0.92, 95% CI 2-sided [0.76 to 1.12]
Statistical Analysis 5: Comparison: cTIV vs eTIV_f; The following hypotheses were tested for A/H3N2 strain as measured by HI cell-culture-derived assay: H0i: log(GMTeTIV_f(i)) - log(GMTcTIV(i)) ≥0.301 ↔ GMTcTIV(i) / GMTeTIV_f(i) ≤0.5 (null hypothesis); H1i: log(GMTeTIV_f(i)) - log(GMTcTIV(i)) <0.301 ↔ GMTcTIV(i) / GMTeTIV_f(i) >0.5 (alternative hypothesis); With: GMTcTIV(i)=GMT for strain i in cTIV group; GMTeTIV_f(i)=GMT for strain i in eTIV_f group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 4]; ANOVA; Ratio of GMT = 0.61, 95% CI 2-sided [0.50 to 0.75]
Statistical Analysis 6: Comparison: cTIV vs eTIV_f; The following hypotheses were tested for B strain as measured by cell-culture-derived assay: H0i: log(GMTeTIV_f(i)) - log(GMTcTIV(i)) ≥0.301 ↔ GMTcTIV(i) / GMTeTIV_f(i) ≤0.5 (null hypothesis); H1i: log(GMTeTIV_f(i)) - log(GMTcTIV(i)) <0.301 ↔ GMTcTIV(i) / GMTeTIV_f(i) >0.5 (alternative hypothesis); With: GMTcTIV(i)=GMT for strain i in cTIV group; GMTeTIV_f(i)=GMT for strain i in eTIV_f group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 4]; ANOVA; Ratio of GMT = 1.31, 95% CI 2-sided [1.09 to 1.57]

2. Secondary Outcome: Geometric Mean Ratio After 1 Dose of Cell-culture-derived Vaccine (cTIV) or Egg-derived Vaccine (eTIV_f), Using the ANOVA Method.
Description: Geometric mean ratio (GMR) of Day 22 / Day 1 geometric mean antibody titers was assessed by egg-derived antigen and cell-derived antigen haemagglutination inhibition (HI) assay.
  The criterion is met according to European (CHMP) guideline if the mean geometric increase GMR (Day22/Day1) in HI antibody titer is > 2.5.
Time Frame: 3 weeks postvaccination (Day 22)
Population: Analysis was done on per protocol set
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | cTIV | eTIV_f
Number analyzed (Participants) | 307 | 303
Ratio
  A/H1N1 (egg-derived assay) | 8.06 [6.64 to 9.8] | 9.65 [7.93 to 12]
  A/H3N2 (egg-derived assay) | 18 [15 to 20] | 25 [21 to 29]
  B (egg-derived assay) | 11 [9.49 to 13] | 9.15 [7.83 to 11]
  A/H1N1 (cell-culture-derived assay) | 9.21 [7.48 to 11] | 10 [8.19 to 12]
  A/H3N2 (cell-culture-derived assay) | 18 [15 to 21] | 22 [18 to 26]
  B (cell-culture-derived assay) | 10 [8.92 to 12] | 7.6 [6.54 to 8.83]

3. Secondary Outcome: Geometric Mean Ratio After 1 Dose of Cell-culture-derived Vaccine (cTIV) or Egg-derived Vaccine (eTIV_f), Using the ANCOVA Method.
Description: as for outcome 2
Time Frame: 3 weeks postvaccination (Day 22)
Population: Analysis was done on per protocol set
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | cTIV | eTIV_f
Number analyzed (Participants) | 307 | 303
Ratio
  A/H1N1 (egg-derived assay) | 7.76 [6.36 to 9.47] | 9.32 [7.64 to 11]
  A/H3N2 (egg-derived assay) | 18 [15 to 21] | 25 [22 to 30]
  B (egg-derived assay) | 11 [9.14 to 13] | 8.86 [7.57 to 10]
  A/H1N1 (cell-culture-derived assay) | 8.76 [7.08 to 11] | 9.64 [7.8 to 12]
  A/H3N2 (cell-culture-derived assay) | 18 [15 to 21] | 22 [19 to 26]
  B (cell-culture-derived assay) | 10 [8.76 to 12] | 7.46 [6.41 to 8.68]

4. Secondary Outcome: Geometric Mean Titers (GMT) Before and After 1 Dose of Cell-culture-derived Vaccine (cTIV) or Egg-derived Vaccine (eTIV_f), Using the ANOVA Method
Description: Antibody titers as assessed by egg-derived antigen and cell-derived antigen haemagglutination inhibition (HI) assay.
Time Frame: 3 weeks postvaccination (Day 22)
Population: Analysis was done on per protocol set
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | cTIV | eTIV_f
Number analyzed (Participants) | 307 | 303
Titer
  A/H1N1 (Day 1) (egg-derived assay) | 32 [27 to 39] | 32 [26 to 38]
  A/H1N1 (Day 22) (egg-derived assay) | 259 [225 to 298] | 306 [265 to 352]
  A/H1N1 (Day 1) (cell-culture-derived assay) | 51 [42 to 62] | 50 [41 to 61]
  A/H1N1 (Day 22) (cell-culture-derived assay) | 468 [407 to 538] | 508 [441 to 585]
  A/H3N2 (Day 1) (egg derived assay) | 10 [9.22 to 12] | 13 [12 to 15]
  A/H3N2 (Day 22) (egg-derived assay) | 181 [157 to 210] | 320 [276 to 370]
  A/H3N2 (Day 1) (cell-culture-derived assay) | 16 [14 to 18] | 21 [19 to 24]
  A/H3N2 (Day 22) (cell-culture-derived assay) | 287 [250 to 331] | 468 [406 to 539]
  B (Day 1) (egg-derived assay) | 16 [14 to 18] | 17 [15 to 20]
  B (Day 22) (egg-derived assay) | 179 [157 to 203] | 157 [138 to 179]
  B (Day 1) (cell-culture-derived assay) | 17 [15 to 19] | 18 [15 to 20]
  B (Day 22) (cell-culture-derived assay) | 176 [155 to 199] | 134 [118 to 153]

5. Secondary Outcome: Percentages of Subjects With Haemagglutination Inhibition (HI) Antibody Titer ≥ 40.
Description: Antibody titers as assessed by egg-derived antigen and cell-derived antigen HI assay.
  This criterion is met according to European (CHMP) guideline if the percentages of subjects achieving HI titers ≥40 is >70%. According to the US Center for Biologics Evaluation and Research (CBER) guideline, the criterion is also met if the lower limit of the 95% CI for percentages of subjects achieving seroprotection (HI antibody titer ≥1:40) is ≥70%.
Time Frame: 3 weeks postvaccination (Day 22)
Population: Analysis was done on per protocol set
Measure: Number (95% Confidence Interval); unit: Percentages
Groups:
- cTIV: Adults 18 to < 50 years of age received one dose of cell- culture-derived trivalent influenza vaccine (cTIV).
Arm/Group | cTIV | eTIV_f
Number analyzed (Participants) | 307 | 303
Percentages
  A/H1N1 (egg-derived assay) | 96 [94 to 98] | 98 [96 to 99]
  A/H3N2 (egg-derived assay) | 91 [87 to 94] | 96 [93 to 98]
  B (egg-derived assay) | 94 [91 to 96] | 93 [89 to 95]
  A/H1N1 (cell-culture-derived assay) | 99 [98 to 100] | 99 [97 to 100]
  A/H3N2 (cell-culture-derived assay) | 98 [95 to 99] | 99 [97 to 100]
  B(cell-culture-derived assay) | 97 [94 to 98] | 91 [88 to 94]

6. Secondary Outcome: Percentages of Subjects With Seroconversion.
Description: As the definition for seroconversion/significant increase from CHMP guideline CPMP/BWP/214/96 corresponds to that of seroconversion from the May 2007 CBER guidance, the analysis of this immunogenicity endpoint is presented as seroconversion. Seroconversion is defined as prevaccination HI titer <10 and postvaccination HI titer ≥40, or prevaccination HI titer ≥10 and a ≥4-fold increase in postvaccination HI antibody titer, on day 22. CBER criterion is met if the lower limit of the 95% CI for percentages of subjects achieving seroconversion for HI antibody (at least a 4-fold rise in HI antibody titer) postvaccination is ≥40%. CHMP criterion is also met if the percentages of subjects achieving seroconversion is >40%.
Time Frame: 3 weeks postvaccination (Day 22)
Population: Analysis was done on per protocol set
Measure: Number (95% Confidence Interval); unit: Percentages
Arm/Group | cTIV | eTIV_f
Number analyzed (Participants) | 307 | 303
Percentages
  A/H1N1 (egg-derived assay) | 62 [57 to 68] | 65 [59 to 70]
  A/H3N2 (egg-derived assay) | 85 [81 to 89] | 92 [88 to 95]
  B (egg-derived assay) | 77 [72 to 81] | 76 [70 to 80]
  A/H1N1 (cell-culture-derived assay) | 62 [56 to 67] | 64 [58 to 69]
  A/H3N2 (cell-culture-derived assay) | 89 [85 to 92] | 90 [87 to 93]
  B(cell-culture-derived assay) | 78 [73 to 83] | 72 [66 to 77]

7. Primary Outcome: Geometric Mean Titers (GMT) After 1 Dose of Cell-culture-derived Vaccine (cTIV) or Egg-derived Vaccine (eTIV_f), Using the ANCOVA Method.
Description: as for outcome 1
Time Frame: 3 weeks postvaccination (Day 22)
Population: Analysis was done on per protocol set
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | cTIV | eTIV_f
Number analyzed (Participants) | 307 | 303
Titer
  A/H1N1 (egg-derived assay) | 263 [229 to 302] | 310 [270 to 355]
  A/H3N2 (egg-derived assay) | 199 [173 to 229] | 316 [275 to 364]
  B (egg-derived assay) | 185 [163 to 210] | 159 [141 to 181]
  A/H1N1 (cell-culture-derived assay) | 478 [417 to 549] | 518 [451 to 595]
  A/H3N2 (cell-culture-derived assay) | 306 [267 to 350] | 444 [388 to 508]
  B (cell-culture-derived assay) | 180 [160 to 203] | 135 [120 to 153]
Statistical Analysis 1: Comparison: cTIV vs eTIV_f; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; Ratio of GMT = 0.85, 95% CI 2-sided [0.70 to 1.03]
Statistical Analysis 2: Comparison: cTIV vs eTIV_f; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; Ratio of GMT = 0.63, 95% CI 2-sided [0.52 to 0.76]
Statistical Analysis 3: Comparison: cTIV vs eTIV_f; [analysis description as in outcome 1, analysis 3]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; Ratio of GMT = 1.16, 95% CI 2-sided [0.98 to 1.38]
Statistical Analysis 4: Comparison: cTIV vs eTIV_f; [analysis description as in outcome 1, analysis 4]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA — To demonstrate non-inferiority of cTIV to eTIV_f the lower limit of the 95% confidence interval (CI) around the ratio of the postvaccination GMTs had to be >0.5; Ratio of GMT = 0.92, 95% CI 2-sided [0.76 to 1.12]
Statistical Analysis 5: Comparison: cTIV vs eTIV_f; [analysis description as in outcome 1, analysis 5]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; Ratio of GMT = 0.69, 95% CI 2-sided [0.57 to 0.83]
Statistical Analysis 6: Comparison: cTIV vs eTIV_f; The following hypotheses were tested for B strain as measured by HI cell-culture-derived assay: H0i: log(GMTeTIV_f(i)) - log(GMTcTIV(i)) ≥0.301 ↔ GMTcTIV(i) / GMTeTIV_f(i) ≤0.5 (null hypothesis); H1i: log(GMTeTIV_f(i)) - log(GMTcTIV(i)) <0.301 ↔ GMTcTIV(i) / GMTeTIV_f(i) >0.5 (alternative hypothesis); With: GMTcTIV(i)=GMT for strain i in cTIV group; GMTeTIV_f(i)=GMT for strain i in eTIV_f group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; Ratio of GMT = 1.33, 95% CI 2-sided [1.13 to 1.58]

8. Secondary Outcome: Number of Subjects Reporting Local and Systemic Reactions
Description: Safety and tolerability of cTIV and eTIV_f postvaccination.
  Difference between demography and safety numbers was due to one misrandomization.
Time Frame: 7 days postvaccination
Population: Analysis was done on safety set
Measure: Number; unit: Subjects
Arm/Group | cTIV | eTIV_f
Number analyzed (Participants) | 309 | 304
Subjects
  Ecchymosis | 12 | 26
  Injection site erythema | 34 | 48
  Injection site induration | 27 | 19
  Injection site swelling | 13 | 16
  Injection site pain | 155 | 169
  Chills | 14 | 26
  Malaise | 76 | 72
  Myalgia | 68 | 73
  Arthralgia | 26 | 28
  Headache | 109 | 121
  Sweating | 15 | 23
  Fatigue | 59 | 67
  Nausea | 31 | 35
  Cough | 26 | 35
  Wheezing | 7 | 9
  Chest tightness | 14 | 11
  Difficulty breathing | 10 | 6
  Sore Throat | 53 | 45
  Facial Edema | 1 | 1
  Red Eye | 3 | 6
  Fever (>=38°C)) | 3 | 3
  Stayed at home due to reaction | 7 | 9
  Analgesic medicine used | 102 | 109

ADVERSE EVENTS:
Time Frame: All Serious adverse events were collected throughout the study period (Day 1 - Day 180). All solicited adverse reactions were collected from Day 1 - Day 7. All unsolicited reactions were collected from Day 8 - Day 180.
Arm/Group | cTIV | eTIV_f
Serious Adverse Events (participants affected / at risk) | 3/309 | 5/304
Other Adverse Events (participants affected / at risk) | 236/309 | 237/304
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | cTIV (N=309) | eTIV_f (N=304)
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 2
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Nasal septal operation (Surgical and medical procedures) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | cTIV (N=309) | eTIV_f (N=304)
Injection site pain (General disorders) | 155 | 169
Headache (Nervous system disorders) | 109 | 121
Malaise (General disorders) | 76 | 72
Myalgia (Musculoskeletal and connective tissue disorders) | 68 | 73
Fatigue (General disorders) | 60 | 67
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 53 | 45
Injection site erythema (General disorders) | 34 | 48
Cough (Respiratory, thoracic and mediastinal disorders) | 26 | 35
Nausea (Gastrointestinal disorders) | 31 | 35
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 | 29
Injection site induration (General disorders) | 27 | 19
Chills (General disorders) | 14 | 26
Injection site haemorrhage (General disorders) | 12 | 26
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 15 | 23
Injection site swelling (General disorders) | 13 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days